CLINICAL TRIAL: NCT03500679
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate Safety and Immunogenicity of the ExPEC4V (JNJ-63871860) Clinical Trial Material After a Single Intramuscular Dose and a Second Dose 6 Months Later in Healthy Subjects Aged 18 Years and Older
Brief Title: A Study to Evaluate Safety and Immunogenicity of the ExPEC4V Clinical Trial Material After a Single Intramuscular Dose and a Second Dose 6 Months Later in Healthy Participants Aged 18 Years and Older
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CR108447; 63871860BAC2003 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2018-04-10; First posted 2018-04-18 (Actual); Results first posted 2019-11-26 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1: ExPEC4V (JNJ-63871860) (Experimental): Participants will receive vaccination of ExPEC4V dose as an intramuscular (IM) injection into deltoid muscle on Days 1 and 181. The ExPEC4V doses contain polysaccharide antigen (4:4:4:8 microgram [mcg]) from the ExPEC4V serotypes O1A, O2, O6A, and O25B.
  Interventions: Biological: ExPEC4V
- Group 2: Placebo (Placebo Comparator): Participants will receive placebo matching to ExPEC4V as an IM injection on Days 1 and 181.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: ExPEC4V — Participants will receive ExPEC4V vaccine as an IM injection on Days 1 and 181.
  Other Names: JNJ-63871860
  Arms: Group 1: ExPEC4V (JNJ-63871860)
Biological: Placebo — Participants will receive placebo as an IM injection on Days 1 and 181.
  Arms: Group 2: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety/reactogenicity of the ExPEC4V clinical trial material (CTM) after the first vaccination and to evaluate the immunogenicity of the ExPEC4V CTM, as measured by the enzyme-linked immunosorbent assay (ELISA), 14 days after the first vaccination (on Day 15).

ELIGIBILITY:
Inclusion Criteria:

* Participants who provides written informed consent and signs the informed consent form (ICF) indicating that he or she understands the purpose, procedures and potential risks and benefits of the study, and is willing to participate in the study
* Participant is medically stable as confirmed by documented medical history, physical examination and vital signs. Participant may have underlying illnesses such as hypertension, diabetes, or ischemic heart disease, as long as their symptoms/signs are medically controlled. If he/she is on medication for a condition, the medication dose must have been stable for at least 12 weeks preceding vaccination
* Participant must have a body mass index (BMI) of less than or equal to (<=)35.0 kilogram per square meter (kg/m^2)
* Contraceptive (birth control) use by woman should be consistent with local regulations regarding the acceptable methods of contraception for participant participating in clinical studies
* All females of childbearing potential must have a negative urine beta-human chorionic gonadotropin (beta-hCG) at pregnancy test on Visit 1 (pre-vaccination) and Visit 4 (prior to the second vaccination)

Exclusion Criteria:

* Participant with contraindication to intramuscular (IM) injections and blood draws, for example, bleeding disorders
* Participant with known allergies, hypersensitivity, or intolerance to ExPEC4V or its excipients
* Participant with abnormal function of the immune system resulting from: a) clinical conditions (for example, autoimmune disease or immunodeficiency); b) chronic or recurrent use of systemic corticosteroids; c) administration of antineoplastic and immunomodulating agents or radiotherapy
* Participant has a history of neoplastic disease (excluding non-melanoma skin cancer or carcinoma in situ of the cervix that was successfully treated) within the past 1 year or a history of any hematological malignancy
* Participant with history of acute polyneuropathy (for example, Guillain-Barre syndrome)
* Participant who has a history of an underlying clinically significant acute or (uncontrolled) chronic medical condition or physical examination findings for which, in the opinion of the investigator, participation would not be in the best interest of the participant (for example, compromise the well-being) or that could prevent, limit, or confound the protocol-specified assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-05-09 (Actual); Primary Completion 2018-11-05 (Actual); Study Completion 2019-06-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (2):
- United States (2):
  - Heartland Clinical Research, Wichita, Kansas
  - VGR & NOCCR - Knoxville, Knoxville, Tennessee

RESULTS

PARTICIPANT FLOW:
Groups:
- ExPEC4V: Participants received a single 0.5 milliliter (mL) dose of ExPEC4V vaccine as an intramuscular (IM) injection into the deltoid muscle on Day 1 and Day 181.
- Placebo: Participants received placebo matching to ExPEC4V as an IM injection into the deltoid muscle on Day 1 and Day 181.
Period: Overall Study
Arm/Group | ExPEC4V | Placebo
Started | 75 | 25
Completed | 66 | 22
Not Completed | 9 | 3
Not completed — Lost to Follow-up | 6 | 3
Not completed — Withdrawal by Subject | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ExPEC4V | Placebo | Total
Number analyzed (Participants) | 75 | 25 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.7 (18.86) | 56.4 (17.56) | 55.9 (18.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 13 | 52
  Male | 36 | 12 | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 1 | 6
  Not Hispanic or Latino | 69 | 23 | 92
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 6 | 2 | 8
  White | 63 | 22 | 85
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 3 | 0 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 6 | 2 | 8
  Hispanic or Latino | 1 | 0 | 1
  Other | 7 | 2 | 9
  White Non-Hispanic | 61 | 21 | 82
Region of Enrollment [Count of Participants; unit: Participants]
  UNITED STATES | 75 | 25 | 100

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Solicited Local Adverse Events (AEs) After First Vaccination
Description: An AE is any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the study vaccine. An AE can therefore be any unfavorable and unintended sign (including an abnormal finding), symptom, or disease temporally associated with the use of a medicinal (investigational or non-investigational) product, whether or not related to that medicinal (investigational or non-investigational) product. Solicited local AEs were precisely defined local events that participants were specifically asked about and which were noted by participants in the diary. Solicited local AEs included injection-site pain/tenderness, injection-site erythema and injection-site swelling/induration.
Time Frame: 14 days after first vaccination (Day 1 to Day 15)
Population: The full analysis set (FAS) included all randomized participants with at least one study vaccine administration documented regardless of the occurrence of protocol deviations.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | ExPEC4V | Placebo
Number analyzed (Participants) | 75 | 25
Percentage of participants | 38.7 [27.64 to 50.62] | 20.0 [6.83 to 40.70]

2. Primary Outcome: Percentage of Participants With Solicited Systemic Adverse Events After First Vaccination
Description: An AE is any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the study vaccine. An AE can therefore be any unfavorable and unintended sign (including an abnormal finding), symptom, or disease temporally associated with the use of a medicinal (investigational or non-investigational) product, whether or not related to that medicinal (investigational or non-investigational) product. Solicited systemic AEs were precisely defined systemic events that participants were specifically asked about and which were noted by participants in the diary. Solicited systemic AEs included fatigue, headache, nausea, myalgia and fever.
Time Frame: 14 days after first vaccination (Day 1 to Day 15)
Population: The FAS included all randomized participants with at least one study vaccine administration documented regardless of the occurrence of protocol deviations.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | ExPEC4V | Placebo
Number analyzed (Participants) | 75 | 25
Percentage of participants | 49.3 [37.58 to 61.14] | 20.0 [6.83 to 40.70]

3. Primary Outcome: Percentage of Participants With Unsolicited Adverse Events After First Vaccination
Description: An AE is any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the study vaccine. An AE can therefore be any unfavorable and unintended sign (including an abnormal finding), symptom, or disease temporally associated with the use of a medicinal (investigational or non-investigational) product, whether or not related to that medicinal (investigational or non-investigational) product. Unsolicited AEs were precisely defined events that participants were not asked about and which were not noted by participants in the diary.
Time Frame: 29 days after first vaccination (Day 1 to Day 30)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | ExPEC4V | Placebo
Number analyzed (Participants) | 75 | 25
Percentage of participants | 30.7 [20.53 to 42.38] | 32.0 [14.95 to 53.50]

4. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs) After First Vaccination
Description: An AE is any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the study vaccine. An AE can therefore be any unfavorable and unintended sign (including an abnormal finding), symptom, or disease temporally associated with the use of a medicinal (investigational or non-investigational) product, whether or not related to that medicinal (investigational or non-investigational) product. An SAE is any AE that results in: death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect and is a suspected transmission of any infectious agent via a medicinal product.
Time Frame: Up to Day 180
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | ExPEC4V | Placebo
Number analyzed (Participants) | 75 | 25
Participants | 1 | 1

5. Primary Outcome: Enzyme-linked Immunosorbent Assay (ELISA) Geometric Mean Titers (GMTs) for Serotypes O1A, O2, O6A and O25B at Day 1
Description: Immunoglobulin G (IgG) antibody levels elicited by the vaccine against each of the 4 vaccine serotypes (serotype O1A, O2, O6A and O25B) were measured by ELISA. GMTs for serotypes O1A, O2, O6A and O25B at Day 1 were reported.
Time Frame: Day 1
Population: The per-protocol immunogenicity (PPI) analysis set consisted of all participants from the FAS excluding those with major protocol deviations expecting to impact the immunogenicity outcomes.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | ExPEC4V | Placebo
Number analyzed (Participants) | 74 | 24
Titer
  Serotype O1A | 3177.8 [2412.54 to 4185.68] | 3113.7 [1910.56 to 5074.63]
  Serotype O2 | 3598.1 [2865.83 to 4517.54] | 4127.3 [2182.46 to 7805.05]
  Serotype O6A | 864.6 [664.08 to 1125.58] | 817.9 [473.94 to 1411.46]
  Serotype O25B | 375.3 [285.25 to 493.69] | 550.8 [288.87 to 1050.27]

6. Primary Outcome: ELISA GMTs for Serotypes O1A, O2, O6A and O25B at Day 15
Description: IgG antibody levels elicited by the vaccine against each of the 4 vaccine serotypes (serotype O1A, O2, O6A and O25B) were measured by ELISA. GMTs for serotypes O1A, O2, O6A and O25B at Day 15 were reported.
Time Frame: Day 15
Population: The PPI analysis set consisted of all participants from the FAS excluding those with major protocol deviations expecting to impact the immunogenicity outcomes. Here 'N' (number of participants analyzed) signifies number of participants evaluable for this outcome measure.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | ExPEC4V | Placebo
Number analyzed (Participants) | 73 | 24
Titer
  Serotype O1A | 17030.3 [13048.22 to 22227.66] | 2838.2 [1749.61 to 4604.01]
  Serotype O2 | 44704.8 [33459.35 to 59729.66] | 3761.6 [2129.94 to 6643.37]
  Serotype O6A | 8206.6 [6241.05 to 10791.06] | 746.2 [444.10 to 1253.75]
  Serotype O25B | 6132.4 [4280.78 to 8784.88] | 467.1 [249.47 to 874.61]

7. Primary Outcome: ELISA Geometric Mean Ratio (GMR) for Serotypes O1A, O2, O6A and O25B at Day 15/Day 1
Description: IgG antibody levels elicited by the vaccine against each of the 4 vaccine serotypes (serotype O1A, O2, O6A and O25B) were measured by ELISA. GMR for serotypes O1A, O2, O6A and O25B (Day 15/Day 1) was reported.
Time Frame: Day 15/Day 1
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | ExPEC4V | Placebo
Number analyzed (Participants) | 73 | 24
Ratio
  Serotype O1A | 5.22 [4.142 to 6.568] | 0.91 [0.799 to 1.040]
  Serotype O2 | 12.06 [9.221 to 15.771] | 0.89 [0.682 to 1.149]
  Serotype O6A | 8.61 [6.515 to 11.379] | 0.94 [0.817 to 1.079]
  Serotype O25B | 12.02 [8.460 to 17.090] | 0.87 [0.658 to 1.159]

8. Primary Outcome: Percentage of Participants With a 2-fold and 4-fold Increase From Baseline in Serum Antibody Titers (ELISA) at Day 15
Description: Percentage of participants with a 2-fold and 4-fold increase from baseline in serum antibody titers as measured by ELISA at Day 15 were reported.
Time Frame: Day 15
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | ExPEC4V | Placebo
Number analyzed (Participants) | 73 | 24
Percentage of participants
  Serotype O1A: ELISA 2-fold | 82.2 [71.47 to 90.16] | 0.0 [0.00 to 14.25]
  Serotype O1A: ELISA 4-fold | 57.5 [45.41 to 69.03] | 0.0 [0.00 to 14.25]
  Serotype O2: ELISA 2-fold | 91.8 [82.96 to 96.92] | 0.0 [0.00 to 14.25]
  Serotype O2: ELISA 4-fold | 83.6 [73.05 to 91.21] | 0.0 [0.00 to 14.25]
  Serotype O6A: ELISA 2-fold | 84.9 [74.64 to 92.23] | 0.0 [0.00 to 14.25]
  Serotype O6A: ELISA 4-fold | 75.3 [63.86 to 84.68] | 0.0 [0.00 to 14.25]
  Serotype O25B: ELISA 2-fold | 89.0 [79.54 to 95.15] | 0.0 [0.00 to 14.25]
  Serotype O25B: ELISA 4-fold | 75.3 [63.86 to 84.68] | 0.0 [0.00 to 14.25]

9. Secondary Outcome: Percentage of Participants With Solicited Local Adverse Events After Second Vaccination
Description: as for outcome 1
Time Frame: 14 days after second vaccination (Day 181 to Day 195)
Population: The FAS included all randomized participants with at least one study vaccine administration documented regardless of the occurrence of protocol deviations. Here 'N' (number of participants analyzed) signifies number of participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | ExPEC4V | Placebo
Number analyzed (Participants) | 68 | 24
Percentage of participants | 45.6 [33.45 to 58.12] | 4.2 [0.11 to 21.12]

10. Secondary Outcome: Percentage of Participants With Solicited Systemic Adverse Events After Second Vaccination
Description: as for outcome 2
Time Frame: 14 days after second vaccination (Day 181 to Day 195)
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | ExPEC4V | Placebo
Number analyzed (Participants) | 68 | 24
Percentage of participants | 48.5 [36.22 to 60.97] | 29.2 [12.62 to 51.09]

11. Secondary Outcome: Percentage of Participants With Unsolicited Adverse Events After Second Vaccination
Description: as for outcome 3
Time Frame: 29 days after second vaccination (Day 181 to Day 210)
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | ExPEC4V | Placebo
Number analyzed (Participants) | 68 | 24
Percentage of participants | 11.8 [5.22 to 21.87] | 8.3 [1.03 to 27.00]

12. Secondary Outcome: Number of Participants With Serious Adverse Events After Second Vaccination
Description: as for outcome 4
Time Frame: Day 181 until Day 360
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | ExPEC4V | Placebo
Number analyzed (Participants) | 68 | 24
Participants | 1 | 0

13. Secondary Outcome: Opsonophagocytic Killing Assay (OPKA) GMTs for Serotypes O1A, O2, O6A and O25B at Days 1 and 15
Description: Specific functional antibacterial antibodies were measured by OPKA. GMTs for serotypes O1A, O2, O6A and O25B at Days 1 and 15 were reported.
Time Frame: Days 1 and 15
Population: The PPI analysis set consisted of all participants from the FAS excluding those with major protocol deviations expecting to impact the immunogenicity outcomes. Here 'n' (number analyzed) signifies number of participants evaluable for specified time points for specified categories.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | ExPEC4V | Placebo
Number analyzed (Participants) | 74 | 24
Titer
  Serotype O1A: Day 1 | 156.8 [131.76 to 186.53] | 173.0 [116.55 to 256.69]
  Serotype O1A: Day 15: number analyzed (Participants) | 73 | 24
  Serotype O1A: Day 15 | 735.6 [535.33 to 1010.75] | 165.3 [111.87 to 244.12]
  Serotype O2: Day 1 | 207.2 [167.79 to 255.74] | 295.0 [179.18 to 485.64]
  Serotype O2: Day 15: number analyzed (Participants) | 73 | 24
  Serotype O2: Day 15 | 2667.3 [1896.34 to 3751.64] | 241.8 [156.39 to 373.80]
  Serotype O6A: Day 1 | 304.8 [229.09 to 405.46] | 380.7 [217.04 to 667.59]
  Serotype O6A: Day 15: number analyzed (Participants) | 73 | 24
  Serotype O6A: Day 15 | 802.4 [632.29 to 1018.16] | 468.5 [241.48 to 908.80]
  Serotype O25B: Day 1 | 68.8 [54.64 to 86.65] | 59.3 [39.08 to 90.08]
  Serotype O25B: Day 15: number analyzed (Participants) | 73 | 24
  Serotype O25B: Day 15 | 188.9 [141.11 to 252.78] | 51.9 [35.59 to 75.63]

14. Secondary Outcome: OPKA GMR for Serotypes O1A, O2, O6A and O25B at Day 15/Day 1
Description: Specific functional antibacterial antibodies were measured by OPKA. GMR for serotypes O1A, O2, O6A and O25B (Day 15/Day 1) was reported.
Time Frame: Day 15/Day 1
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | ExPEC4V | Placebo
Number analyzed (Participants) | 73 | 24
Ratio
  Serotype O1A | 3.47 [2.687 to 4.479] | 0.98 [0.959 to 1.009]
  Serotype O2 | 10.78 [7.943 to 14.631] | 0.84 [0.629 to 1.132]
  Serotype O6A | 2.49 [1.989 to 3.120] | 1.23 [0.834 to 1.816]
  Serotype O25B | 2.37 [1.892 to 2.976] | 0.87 [0.739 to 1.034]

15. Secondary Outcome: Percentage of Participants With a 2-fold and 4-fold Increase From Baseline in Serum Antibody Titers (OPKA) at Day 15
Description: Percentage of participants with a 2-fold and 4-fold increase from baseline in serum antibody titers as measured by OPKA at Day 15 were reported.
Time Frame: Day 15
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | ExPEC4V | Placebo
Number analyzed (Participants) | 73 | 24
Percentage of participants
  Serotype O1A: OPKA 2-fold | 64.4 [52.31 to 75.25] | 0.0 [0.00 to 14.25]
  Serotype O1A: OPKA 4-fold | 41.1 [29.71 to 53.23] | 0.0 [0.00 to 14.25]
  Serotype O2: OPKA 2-fold | 86.3 [76.25 to 93.23] | 0.0 [0.00 to 14.25]
  Serotype O2: OPKA 4-fold | 72.6 [60.91 to 82.39] | 0.0 [0.00 to 14.25]
  Serotype O6A: OPKA 2-fold | 46.6 [34.80 to 58.63] | 8.3 [1.03 to 27.00]
  Serotype O6A: OPKA 4-fold | 23.3 [14.19 to 34.65] | 8.3 [1.03 to 27.00]
  Serotype O25B: OPKA 2-fold | 46.6 [34.80 to 58.63] | 0.0 [0.00 to 14.25]
  Serotype O25B: OPKA 4-fold | 21.9 [13.08 to 33.14] | 0.0 [0.00 to 14.25]

16. Secondary Outcome: ELISA GMTs for Serotypes O1A, O2, O6A, O25B at Days 181 and 195
Description: IgG antibody levels elicited by the vaccine against each of the 4 vaccine serotypes (serotype O1A, O2, O6A, O25B) were measured by ELISA. GMTs for serotypes O1A, O2, O6A and O25B at Days 181 and 195 were reported.
Time Frame: Days 181 and 195
Population: Analysis population included PPI analysis set. Here 'N' (number of participants analyzed) signifies number of participants evaluable for this outcome measure and 'n' (number analyzed) signifies number of participants evaluable for specified time points for specified categories.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | ExPEC4V | Placebo
Number analyzed (Participants) | 67 | 24
Titer
  Serotype O1A: Day 181 | 10445.0 [7931.32 to 13755.33] | 3245.8 [1968.83 to 5351.07]
  Serotype O1A: Day 195: number analyzed (Participants) | 64 | 24
  Serotype O1A: Day 195 | 14347.1 [10821.68 to 19020.91] | 3214.6 [1987.00 to 5200.52]
  Serotype O2: Day 181 | 27748.0 [20310.07 to 37909.76] | 5187.8 [2866.53 to 9388.63]
  Serotype O2: Day 195: number analyzed (Participants) | 64 | 24
  Serotype O2: Day 195 | 34841.7 [26020.58 to 46653.16] | 5252.6 [2980.81 to 9255.68]
  Serotype O6A: Day 181 | 4658.9 [3592.36 to 6042.17] | 1014.4 [596.31 to 1725.64]
  Serotype O6A: Day 195: number analyzed (Participants) | 64 | 24
  Serotype O6A: Day 195 | 7716.8 [6034.01 to 9868.80] | 1057.8 [635.59 to 1760.42]
  Serotype O25B: Day 181 | 2089.0 [1488.57 to 2931.67] | 541.1 [286.50 to 1021.82]
  Serotype O25B: Day 195: number analyzed (Participants) | 64 | 24
  Serotype O25B: Day 195 | 4212.3 [3010.69 to 5893.61] | 532.1 [281.44 to 1005.88]

17. Secondary Outcome: ELISA GMR for Serotype O1A, O2, O6A and O25B at Day 181/Day 1 and Day 195/Day 1
Description: IgG antibody levels elicited by the vaccine against each of the 4 vaccine serotypes (serotype O1A, O2, O6A and O25B) were measured by ELISA. GMR for serotypes O1A, O2, O6A and O25B (Day 181/Day 1 and Day 195/Day 1) was reported.
Time Frame: Day 181/Day 1 and Day 195/Day 1
Population: as for outcome 16
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | ExPEC4V | Placebo
Number analyzed (Participants) | 67 | 24
Ratio
  Serotype O1A: Day 181/Day 1 | 3.30 [2.694 to 4.046] | 1.04 [0.915 to 1.188]
  Serotype O1A: Day 195/Day 1: number analyzed (Participants) | 64 | 24
  Serotype O1A: Day 195/Day 1 | 4.42 [3.571 to 5.466] | 1.03 [0.914 to 1.166]
  Serotype O2: Day 181/Day 1 | 7.78 [5.965 to 10.154] | 1.22 [1.097 to 1.359]
  Serotype O2: Day 195/Day 1: number analyzed (Participants) | 64 | 24
  Serotype O2: Day 195/Day 1 | 9.88 [7.608 to 12.832] | 1.20 [1.085 to 1.330]
  Serotype O6A: Day 181/Day 1 | 4.85 [3.879 to 6.070] | 1.20 [0.999 to 1.453]
  Serotype O6A: Day 195/Day 1: number analyzed (Participants) | 64 | 24
  Serotype O6A: Day 195/Day 1 | 8.22 [6.631 to 10.183] | 1.22 [1.018 to 1.464]
  Serotype O25B: Day 181/Day 1 | 4.39 [3.229 to 5.966] | 0.98 [0.853 to 1.132]
  Serotype O25B: Day 195/Day 1: number analyzed (Participants) | 64 | 24
  Serotype O25B: Day 195/Day 1 | 8.51 [6.153 to 11.773] | 0.97 [0.867 to 1.076]

18. Secondary Outcome: Percentage of Participants With a 2-fold and 4-fold Increase From Baseline in Serum Antibody Titers (ELISA) at Days 181 and 195
Description: Percentage of participants with a 2-fold and 4-fold increase from baseline in serum antibody titers as measured by ELISA at Days 181 and 195 were reported.
Time Frame: Days 181 and 195
Population: as for outcome 16
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | ExPEC4V | Placebo
Number analyzed (Participants) | 67 | 24
Percentage of participants
  Serotype O1A: ELISA 2-fold: Day 181 | 64.2 [51.53 to 75.53] | 4.2 [0.11 to 21.12]
  Serotype O1A: ELISA 2-fold: Day 195: number analyzed (Participants) | 64 | 24
  Serotype O1A: ELISA 2-fold: Day 195 | 81.3 [69.54 to 89.92] | 0.0 [0.00 to 14.25]
  Serotype O1A: ELISA 4-fold: Day 181 | 37.3 [25.80 to 49.99] | 0.00 [0.00 to 14.25]
  Serotype O1A: ELISA 4-fold: Day 195: number analyzed (Participants) | 64 | 24
  Serotype O1A: ELISA 4-fold: Day 195 | 57.8 [44.82 to 70.06] | 0.0 [0.00 to 14.25]
  Serotype O2: ELISA 2-fold: Day 181 | 85.1 [74.26 to 92.60] | 0.0 [0.00 to 14.25]
  Serotype O2: ELISA 2-fold: Day 195: number analyzed (Participants) | 64 | 24
  Serotype O2: ELISA 2-fold: Day 195 | 95.3 [86.91 to 99.02] | 0.0 [0.00 to 14.25]
  Serotype O2: ELISA 4-fold: Day 181 | 73.1 [60.90 to 83.24] | 0.0 [0.00 to 14.25]
  Serotype O2: ELISA 4-fold: Day 195: number analyzed (Participants) | 64 | 24
  Serotype O2: ELISA 4-fold: Day 195 | 82.8 [71.32 to 91.10] | 0.0 [0.0 to 14.25]
  Serotype O6A: ELISA 2-fold: Day 181 | 79.1 [67.43 to 88.08] | 8.3 [1.03 to 27.00]
  Serotype O6A: ELISA 2-fold: Day 195: number analyzed (Participants) | 64 | 24
  Serotype O6A: ELISA 2-fold: Day 195 | 95.3 [86.91 to 99.02] | 8.3 [1.03 to 27.00]
  Serotype O6A: ELISA 4-fold: Day 181 | 59.7 [47.00 to 71.51] | 4.2 [0.11 to 21.12]
  Serotype O6A: ELISA 4-fold: Day 195: number analyzed (Participants) | 64 | 24
  Serotype O6A: ELISA 4-fold: Day 195 | 78.1 [66.03 to 87.49] | 4.2 [0.11 to 21.12]
  Serotype O25B: ELISA 2-fold: Day 181 | 65.7 [53.06 to 76.85] | 0.0 [0.00 to 14.25]
  Serotype O25B: ELISA 2-fold: Day 195: number analyzed (Participants) | 64 | 24
  Serotype O25B: ELISA 2-fold: Day 195 | 85.9 [74.98 to 93.36] | 0.0 [0.00 to 14.25]
  Serotype O25B: ELISA 4-fold: Day 181 | 43.3 [31.22 to 55.96] | 0.0 [0.00 to 14.25]
  Serotype O25B: ELISA 4-fold: Day 195: number analyzed (Participants) | 64 | 24
  Serotype O25B: ELISA 4-fold: Day 195 | 67.2 [54.31 to 78.41] | 0.0 [0.00 to 14.25]

19. Secondary Outcome: OPKA GMTs for Serotypes O1A, O2, O6A and O25B at Days 181 and 195
Description: Specific functional antibacterial antibodies were measured by OPKA. GMTs for serotypes O1A, O2, O6A and O25B at Days 181 and 195 were reported.
Time Frame: Days 181 and 195
Population: as for outcome 16
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | ExPEC4V | Placebo
Number analyzed (Participants) | 67 | 24
Titer
  Serotype O1A: Day 181 | 313.9 [234.11 to 420.81] | 153.1 [104.05 to 225.12]
  Serotype O1A: Day 195: number analyzed (Participants) | 64 | 24
  Serotype O1A: Day 195 | 431.1 [317.40 to 585.52] | 151.3 [103.91 to 220.32]
  Serotype O2: Day 181 | 1145.3 [800.61 to 1638.42] | 228.9 [142.75 to 367.06]
  Serotype O2: Day 195: number analyzed (Participants) | 64 | 24
  Serotype O2: Day 195 | 1366.2 [981.63 to 1901.43] | 220.5 [138.74 to 350.58]
  Serotype O6A: Day 181 | 372.3 [298.21 to 464.89] | 324.0 [202.09 to 519.30]
  Serotype O6A: Day 195: number analyzed (Participants) | 64 | 24
  Serotype O6A: Day 195 | 555.8 [459.19 to 672.64] | 328.0 [200.93 to 535.47]
  Serotype O25B: Day 181 | 96.6 [75.68 to 123.23] | 57.3 [37.78 to 87.00]
  Serotype O25B: Day 195: number analyzed (Participants) | 64 | 24
  Serotype O25B: Day 195 | 145.2 [108.32 to 194.65] | 55.0 [35.96 to 84.27]

20. Secondary Outcome: OPKA GMR for Serotype O1A, O2, O6A and O25B at Day 181/Day 1 and Day 195/Day 1
Description: Specific functional antibacterial antibodies were measured by OPKA. GMR for serotypes O1A, O2, O6A and O25B at Day 181/Day 1 and Day 195/Day 1 were reported.
Time Frame: Day 181/Day 1 and Day 195/Day 1
Population: as for outcome 16
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | ExPEC4V | Placebo
Number analyzed (Participants) | 67 | 24
Ratio
  Serotype O1A: Day 181/Day 1 | 1.77 [1.473 to 2.139] | 0.94 [0.842 to 1.043]
  Serotype O1A: Day 195/Day 1: number analyzed (Participants) | 64 | 24
  Serotype O1A: Day 195/Day 1 | 2.27 [1.849 to 2.798] | 0.93 [0.838 to 1.025]
  Serotype O2: Day 181/Day 1 | 4.98 [3.703 to 6.704] | 0.82 [0.717 to 0.943]
  Serotype O2: Day 195/Day 1: number analyzed (Participants) | 64 | 24
  Serotype O2: Day 195/Day 1 | 5.97 [4.576 to 7.785] | 0.79 [0.694 to 0.905]
  Serotype O6A: Day 181/Day 1 | 1.25 [1.022 to 1.522] | 0.83 [0.660 to 1.036]
  Serotype O6A: Day 195/Day 1: number analyzed (Participants) | 64 | 24
  Serotype O6A: Day 195/Day 1 | 1.77 [1.403 to 2.234] | 0.84 [0.676 to 1.037]
  Serotype O25B: Day 181/Day 1 | 1.30 [1.142 to 1.483] | 0.99 [0.870 to 1.137]
  Serotype O25B: Day 195/Day 1: number analyzed (Participants) | 64 | 24
  Serotype O25B: Day 195/Day 1 | 1.89 [1.555 to 2.297] | 0.95 [0.829 to 1.101]

21. Secondary Outcome: Percentage of Participants With a 2-fold and 4-fold Increase From Baseline in Serum Antibody Titers (OPKA) at Days 181 and 195
Description: Percentage of participants with a 2-fold and 4-fold increase from baseline in serum antibody titers as measured by OPKA at Days 181 and 195 were reported.
Time Frame: Days 181 and 195
Population: as for outcome 16
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | ExPEC4V | Placebo
Number analyzed (Participants) | 67 | 24
Percentage of participants
  Serotype O1A: OPKA 2-fold: Day 181 | 38.8 [27.14 to 51.50] | 0.0 [0.00 to 14.25]
  Serotype O1A: OPKA 2-fold: Day 195: number analyzed (Participants) | 64 | 24
  Serotype O1A: OPKA 2-fold: Day 195 | 54.7 [41.75 to 67.18] | 0.0 [0.00 to 14.25]
  Serotype O1A: OPKA 4-fold: Day 181 | 14.9 [7.40 to 25.74] | 0.0 [0.00 to 14.25]
  Serotype O1A: OPKA 4-fold: Day 195: number analyzed (Participants) | 64 | 24
  Serotype O1A: OPKA 4-fold: Day 195 | 31.3 [20.24 to 44.06] | 0.0 [0.00 to 14.25]
  Serotype O2: OPKA 2-fold: Day 181 | 76.1 [64.14 to 85.69] | 0.0 [0.00 to 14.25]
  Serotype O2: OPKA 2-fold: Day 195: number analyzed (Participants) | 64 | 24
  Serotype O2: OPKA 2-fold: Day 195 | 84.4 [73.14 to 92.24] | 0.0 [0.00 to 14.25]
  Serotype O2: OPKA 4-fold: Day 181 | 58.2 [45.52 to 70.15] | 0.0 [0.00 to 14.25]
  Serotype O2: OPKA 4-fold: Day 195: number analyzed (Participants) | 64 | 24
  Serotype O2: OPKA 4-fold: Day 195 | 62.5 [49.51 to 74.30] | 0.0 [0.00 to 14.25]
  Serotype O6A: OPKA 2-fold: Day 181 | 20.9 [11.92 to 32.57] | 0.0 [0.00 to 14.25]
  Serotype O6A: OPKA 2-fold: Day 195: number analyzed (Participants) | 64 | 24
  Serotype O6A: OPKA 2-fold: Day 195 | 34.4 [22.95 to 47.30] | 0.0 [0.00 to 14.25]
  Serotype O6A: OPKA 4-fold: Day 181 | 9.0 [3.36 to 18.48] | 0.0 [0.00 to 14.25]
  Serotype O6A: OPKA 4-fold: Day 195: number analyzed (Participants) | 64 | 24
  Serotype O6A: OPKA 4-fold: Day 195 | 15.6 [7.76 to 26.86] | 0.0 [0.00 to 14.25]
  Serotype O25B: OPKA 2-fold: Day 181 | 14.9 [7.40 to 25.74] | 0.0 [0.00 to 14.25]
  Serotype O25B: OPKA 2-fold: Day 195: number analyzed (Participants) | 64 | 24
  Serotype O25B: OPKA 2-fold: Day 195 | 37.5 [25.70 to 50.49] | 0.0 [0.00 to 14.25]
  Serotype O25B: OPKA 4-fold: Day 181 | 4.5 [0.93 to 12.53] | 0.0 [0.00 to 14.25]
  Serotype O25B: OPKA 4-fold: Day 195: number analyzed (Participants) | 64 | 24
  Serotype O25B: OPKA 4-fold: Day 195 | 17.2 [8.90 to 28.68] | 0.0 [0.00 to 14.25]

ADVERSE EVENTS:
Time Frame: Up to Day 360
Description: The full analysis set (FAS) included all randomized participants with at least one study vaccine administration documented regardless of the occurrence of protocol deviations.
Arm/Group | ExPEC4V | Placebo
All-Cause Mortality (participants affected / at risk) | 0/75 | 0/25
Serious Adverse Events (participants affected / at risk) | 2/75 | 1/25
Other Adverse Events (participants affected / at risk) | 54/75 | 17/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ExPEC4V (N=75) | Placebo (N=25)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Deep Vein Thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ExPEC4V (N=75) | Placebo (N=25)
Bradycardia (Cardiac disorders) | 8 | 1
Nausea (Gastrointestinal disorders) | 17 | 4
Erythema (General disorders) | 3 | 0
Fatigue (General disorders) | 33 | 4
Pain/Tenderness (General disorders) | 36 | 6
Herpes Zoster (Infections and infestations) | 1 | 1
Blood Pressure Diastolic Increased (Investigations) | 2 | 1
Blood Pressure Systolic Increased (Investigations) | 5 | 2
Respiratory Rate Increased (Investigations) | 4 | 1
Gout (Metabolism and nutrition disorders) | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 33 | 7
Headache (Nervous system disorders) | 29 | 5
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Diastolic Hypertension (Vascular disorders) | 0 | 3
Systolic Hypertension (Vascular disorders) | 2 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2017-12-19): https://cdn.clinicaltrials.gov/large-docs/79/NCT03500679/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-22): https://cdn.clinicaltrials.gov/large-docs/79/NCT03500679/SAP_001.pdf